CLINICAL TRIAL: NCT06269406
Title: A Combination of Ibuprofen With Curcumin Covered With Liquorice Root Supplementation in the Management of Postoperative Dental Pain in Adults, Randomized, Double- Blind, Parallel-Group, Placebo-Controlled Study
Brief Title: A Combination of Ibuprofen With Curcumin Covered With Liquorice Root Supplementation in the Management of Postoperative Dental Pain in Adults
Acronym: ICLID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: NMSI DENTMASTER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW008
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Dental Pain
Keywords: Postoperative Dental Pain; Curcumin and Licorice Root; Ibuprofen; Anti-inflammatory Properties; molars
MeSH Terms: conditions — Toothache | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group ibuprofen 400 and Curcumin (Experimental)
  Interventions: Dietary Supplement: ibuprofen 400 mg in combination with Curcumin covered with liquorice root 100 mg
- Intervention Group ibuprofen 200 and Curcumin (Experimental)
  Interventions: Dietary Supplement: ibuprofen 200 mg in combination with Curcumin covered with liquorice root 100 mg
- Intervention Group ibuprofen 400 and placebo (Placebo Comparator)
  Interventions: Other: The combination of ibuprofen 400 mg and placebo in patients after 2-4 molars procedure

INTERVENTIONS:
Dietary Supplement: ibuprofen 400 mg in combination with Curcumin covered with liquorice root 100 mg — The combination of ibuprofen 400 mg and Curcumin covered with liquorice root 100 mg in patients after 2-4 molars procedure
  Arms: Intervention Group ibuprofen 400 and Curcumin
Dietary Supplement: ibuprofen 200 mg in combination with Curcumin covered with liquorice root 100 mg — The combination of ibuprofen 200 mg and Curcumin covered with liquorice root 100 mg in patients after 2-4 molars procedure
  Arms: Intervention Group ibuprofen 200 and Curcumin
Other: The combination of ibuprofen 400 mg and placebo in patients after 2-4 molars procedure — The combination of ibuprofen 400 mg and placebo 100 mg in patients after 2-4 molars procedure
  Arms: Intervention Group ibuprofen 400 and placebo

SUMMARY:
Dental pain, a common issue in stomatology, requires a multifaceted treatment approach. This study explores the efficacy of combining Ibuprofen with curcumin and liquorice root supplements for managing postoperative dental pain. Curcumin, known for its antioxidant and anti-inflammatory properties, along with liquorice root, may enhance pain relief beyond conventional NSAIDs like Ibuprofen. This randomized, double-blind, placebo-controlled trial aims to evaluate the safety and effectiveness of this combination therapy in adults undergoing the removal of impacted third molars. Participants, aged 18-85, were divided into groups receiving different doses of Ibuprofen and curcumin with liquorice root, compared to a control group receiving Ibuprofen and placebo. The primary outcome is the sum of pain intensity differences over 8 hours, with secondary outcomes including total pain relief and the occurrence of any adverse events. The anticipated sample size, considering a 20% dropout rate, is 264 participants, ensuring the study is powered to detect significant differences in pain management efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Removal of 2 to 4 impacted third molars

Exclusion Criteria:

* Pregnancy or breastfeeding
* Ibuprofen contraindications.
* Allergy to any of the intervention components.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Sum of pain intensity differences (SPID), SPID on the visual analog score VAS (points) | 8 hours

SECONDARY OUTCOMES:
Total pain relief (TOTPAR) % | 8 hours
Time to pain half pain gone (in minutes) | 8 hours
Duration of pain half gone (in minutes) | 8 hours
Any adverse events (facial swelling, nausea, vomiting, headache) (%) | 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Nmsi Dentmaster, Novosibirsk, Novosibirsk Oblast, Russia